CLINICAL TRIAL: NCT00965445
Title: The Comparison of Oxidative Stress Between Inhalation Anesthetics
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Other Study IDs: CGMH-IRB-96-0019B; CGMH-IRB-96-0019B
Record Dates: First submitted 2009-08-23; First posted 2009-08-25 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Oxidative Stress; Cardiac Surgery
Keywords: isoprostanes; mass spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — thirty milliliters of urine was collected from urine bag of patients at the following times: baseline before anesthesia, 30 minutes before cardiopulmonary bypass, during cardiopulmonary bypass, after the end of cardiopulmonary bypass.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cardiac surgery with CPB

SUMMARY:
Oxidative stress is an unavoidable event during cardiac surgery. Isoprostanes have been demonstrated to be a reliable biomarker for the evaluation of oxidative stress in vivo.The aims of this study are(1)to develop an accurate liquid chromatography-tandem mass spectrometry methods for the detection of urinary isoprostane isomers in samples collected from healthy volunteers(for method quality control) and patients receiving a cardiac surgery (2)to investigate the change of isoprostanes after cardiopulmonary bypass(CPB) (3)to investigate the effect of different anesthetics on isoprostanes.

DETAILED DESCRIPTION:
Enhanced production of oxygen free radicals can lead to the generation of oxidative stress, which is harmful to human tissue and organs. Reactive oxygen species are released abruptly during some surgical procedures, and they are the major causes of ischemia-reperfusion injuries.Isoprostanes have been demonstrated to be a reliable biomarker for the evaluation of oxidative stress in vivo. Therefore, accurately monitoring and avoiding the occurrence of oxidative stress during surgery is an important clinical issue.

Isoprostanes are a series of prostaglandin-like compounds produced by non-enzymatic peroxidation of arachidonic acid.The aims of this study are(1)to develop an accurate liquid chromatography-tandem mass spectrometry methods for the detection of urinary isoprostane isomers in samples collected from patients receiving a cardiac surgery (2)to investigate the change of isoprostanes after cardiopulmonary bypass (3)to investigate the effect of different anesthetics on isoprostanes during surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving cardiac valve surgery in ASA II-III physical status

Exclusion Criteria:

* trauma, infection, low ejection fraction (less than 25%), liver cirrhosis, or acute renal failure, and emergency surgery

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients receiving cardiac valve surgery in Taipei Change Gung Memorial Hospital will be invited to participate this study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
isoprostanes isomer as marker of oxidative stress | one day

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hui Teng, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Dept. of Anesthesiology, Chang Gung Memorial Hospital, Taipei, Taiwan